CLINICAL TRIAL: NCT07304570
Title: Enhancing Clinical Presence and Decision-Making in Neurosurgical Clerkships: A Hybrid Model Integrating Virtual Reality and Live-Streamed Encounters
Brief Title: VR-Live Hybrid Neurosurgery Clerkship:Boosting Neurosurgical Presence & Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WestChinaH-HX-2025-03
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Telemedicine
Keywords: Neurosurgical education; live-streaming; clerkship training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: VR Simulation (15 hours)+Live-Streamed Neurosurgical Procedures (20 hours)+Live-Streamed Neurocritical Care Rounds (5 hours)
- Control group (No Intervention): * Pre-recorded neurosurgical videos (20 hours): Matched case types from the Neurosurgical Education and Training Resource (NETR) library, with voiceover but no interactivity.
  * Textbook/journal readings (15 hours): Chapters from Neurosurgery: The Essential Guide and articles from Journal of Neurosurgical Education (aligned with case content).
  * Asynchronous case discussions (5 hours): Text-based forums on the institution's LMS, moderated by faculty (48-hour response window).

INTERVENTIONS:
Other: VR Simulation (15 hours)+Live-Streamed Neurosurgical Procedures (20 hours)+Live-Streamed Neurocritical Care Rounds (5 hours) — 1. VR Simulation (15 hours): Customized modules on the NeuroVR Platform (validated for neurosurgical education):
     * Neuroanatomy (5 hours): 3D interactive models of cerebral cortex, brainstem, cranial nerves, and spinal cord (with vascular/meningeal overlays).
     * Procedural skills (10 hours): Craniotomy basics, ventriculostomy, lumbar puncture, and spine decompression-with real-time feedback on instrument handling and anatomical precision.
  2. Live-Streamed Neurosurgical Procedures (20 hours): 18 diverse cases (brain tumor resection [n=6], spine fusion [n=5], aneurysm clipping [n=3], epilepsy surgery [n=4]) via HIPAA-compliant Zoom for Healthcare. Each session included:
     * Pre-procedure briefing (anatomical landmarks, surgical goals).
     * Intraoperative expert commentary (neurosurgeon + neuroanesthesiologist).
     * Real-time Q&A (focused on neurocritical decision-making: e.g., "How do you adjust resection for eloquent cortex mapping?").
  3. Live-Streamed Neurocritical Care Rounds (5 hours): Week
  Arms: Intervention Group

SUMMARY:
The goal of this randomized controlled trial was to learn whether a hybrid telemedicine curriculum that combines virtual-reality (VR) simulation with interactive live-streamed neurosurgical cases improves neurosurgical intentionality and clinical decision-making in fourth-year medical students whose clerkships were disrupted by COVID-19. It also assessed technical skills, theoretical knowledge, and student experience. The main questions it aimed to answer were:

Does the 4-week hybrid model (VR + live cases) produce greater gains in neurosurgical intentionality and decision-making than traditional online videos and readings? Does the hybrid model improve VR technical skill performance and student satisfaction without harming theoretical knowledge? Researchers randomized 112 students 1:1 to the hybrid intervention (15 h VR neuroanatomy/procedures + 20 h live-streamed surgeries/ICU rounds + real-time Q&A) or a time-matched control group (pre-recorded videos, textbook readings, asynchronous forums).

Participants in both groups:

Completed 40 hours of remote content over 4 weeks Were tested at baseline and post-course on intentionality (modified Zwisch scale), decision-making (neurosurgery-specific SCT), 50-item MCQ knowledge, and VR proficiency metrics Joined focus groups and rated satisfaction on a 5-point Likert scale

ELIGIBILITY:
Inclusion Criteria:

1. Fourth-year medical students assigned to the neurosurgical clerkship rotation
2. Able to participate fully in remote learning (stable internet and VR-headset compatible computer)
3. Provided written informed consent

Exclusion Criteria:

1. Had already completed a prior neurosurgical elective
2. Lacked reliable internet access or hardware required for VR/live-streaming
3. Declined to consent or unable to complete the 4-week curriculum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Neurosurgical Intentionality | 4 weeks
  Neurosurgical Intentionality: Intervention group post-intervention scores were compared with controls, the higer the score, the better the outcome
Clinical decision-making score | 4 weeks
  Clinical Decision-Making Score Range: 24-120 points (5-point Likert, 24 items)
  Levels:
  24-48 = low 49-84 = moderate 85-120 = high The higher the score, the better the outcome

SECONDARY OUTCOMES:
Theoretical Knowledge | 4 weeks
  These comprised of theoretical knowledge with 50-item multiple-choice-questions (MCQ) exam on neuroanatomy, pathology, and surgical indications ,the higer the score, the better the outcome
Technical Skill Performance score | 4 weeks
  Technical Skill Performance with VR proficiency metrics such as time to completion, anatomical accuracy, and instrument error rate from NeuroVR's built-in assessment tool. The higer the score,the better the outcome
Student experience score | 4 weeks
  Student experience using semi-structured focus groups such as 6 groups of 8-10 students/group and reflective journals, analyzed via Braun & Clarke's thematic analysis ; and satisfaction using 12-item Likert scale (1=strongly dissatisfied to 5=strongly satisfied) measuring curriculum relevance, engagement, and skill development. The higher the score, the better the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Protocol
Supporting Information: Study Protocol, ICF